CLINICAL TRIAL: NCT02095223
Title: Effect of Electromyographic Biofeedback on Quadriceps Neuromuscular Function
Brief Title: Effect of Electromyographic Biofeedback on Quadriceps Neuromuscular Function in Patients With Quadriceps Inhibition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with participant recruitment.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Christopher Kuenze, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130868
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Knee Injuries
Keywords: Knee injury; Meniscus injury; Anterior cruciate ligament injury; Knee ligament injury
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electromyographic Biofeedback Group (Experimental): Participants in the electromyographic biofeedback supplemented exercise will be instructed on correct setup and use of the electromyographic biofeedback unit. Electromyographic biofeedback will be used during all exercises throughout the course of the study for this group. Participants in will be instructed on a 14 day exercise protocol on the day of enrollment. The protocol is comprised of 4 exercises focused on both non-weight bearing and weight bearing quadriceps strengthening. A compliance log will be given to each participant and will be reviewed at each supervised exercise session and at the final study visit. Participants will be instructed to discontinue exercise and contact the principle investigator if they experience knee pain due to the intervention.
  Interventions: Device: Electromyographic Biofeedback; Behavioral: Traditional Exercise
- Traditional Exercise Group (Active Comparator): Participants in will be instructed on a 14 day exercise protocol on the day of enrollment. The protocol is comprised of 4 exercises focused on both non-weight bearing and weight bearing quadriceps strengthening. A compliance log will be given to each participant and will be reviewed at each supervised exercise session and at the final study visit. Participants will be instructed to discontinue exercise and contact the principle investigator if they experience knee pain due to the intervention.
  Interventions: Behavioral: Traditional Exercise

INTERVENTIONS:
Device: Electromyographic Biofeedback — Electromyographic biofeedback is a device that enables a patient or clinician to measure the intensity of a muscle contraction using electrodes placed on the skin over a muscle of interest. In this study, participants in the electromyographic biofeedback supplemented exercise will also be instructed on correct setup and use of the electromyographic biofeedback unit. These instructions will focus on correct placement of the electromyographic recording electrodes over quadriceps muscle as well as correct tuning of the feedback threshold for each exercise to maximize the benefit of the intervention. Electromyographic biofeedback will be used during all exercises throughout the course of the study for this group.
  Other Names: Device Name: MyoTrac Biofeedback Unit; System#: SA4000P/SA4001P; System Name: Myotrac EMG Biofeedback System
  Arms: Electromyographic Biofeedback Group
Behavioral: Traditional Exercise — All participants will be asked to complete 3 set of 10 repetitions of isometric quadriceps contractions with a 15 second hold time, supine straight leg raises, body weight squatting, and body weight lunges daily. Participants will be required to complete the single limb exercises on the previously injured limb only.

SUMMARY:
Muscle inhibition prevents optimal contraction of the quadriceps muscle due to changes in the nervous system after knee joint injury. Current treatments for muscle inhibition at this time include knee joint cryotherapy and electric stimulation prior to exercise. These treatments, in addition to strengthening exercises, have shown improvements in the quality and strength of muscle contractions however, they have a short window of effectiveness. Electromyographic Biofeedback is proven to be useful in improving quadriceps strength but the mechanism of action remains somewhat unclear. Therefore, the purpose of this investigation is to compare the effectiveness of electromyographic biofeedback supplemented exercise when compared to traditional exercise on quadriceps muscle function in individuals with a history of knee injury and current evidence of quadriceps inhibition. We hypothesize that 14 days of electromyographic biofeedback supplemented exercise will lead to larger gains in quadriceps activation when compared to traditional exercise.

Thirty 18-40 year old participants with a history of knee injury and current evidence of quadriceps muscle inhibition will be enrolled in this single blind randomized controlled trial. Participants will provide written consent prior to all study procedures. Following enrollment, participants will be asked complete questionnaires related to knee related function, current levels of pain, and current activity level followed by completion of baseline measurements.

1. We will use the superimposed burst technique to quadriceps muscle activation.
2. We will measure the Hoffmann reflex response of the quadriceps with surface electromyography. We will measure this signal with surface electromyography electrodes that record the activity of the quadriceps muscle through the skin.

Participants in both groups will be instructed on a 14 day home exercise protocol on the day of enrollment. The protocol is comprised of 4 exercises focused on both non-weight bearing and weight bearing quadriceps strengthening. Compliance will be monitored via a daily exercise diary which will be collected at the end of the study protocol.

Quadriceps central activation ratio, active motor threshold and Hoffmann reflex will be reported descriptively. Pre-intervention and post 14 day intervention quadriceps central activation ratio and Hoffmann reflex will be compared between traditional exercise and Biofeedback supplemented exercise

DETAILED DESCRIPTION:
Screening Subjects will be asked to complete a brief questionnaire about their lower extremity, which will be used to determine if they exhibit any of the exclusionary criteria (administered by the Study Coordinator). This will include past medical history, headache/ migraine history, and any drugs/medications they are currently taking (which might influence the excitability threshold Hoffman reflex (H-reflex) measurement or central activation ratio). Subjects will also undergo quadriceps central activation ratio testing to determine the level of quadriceps inhibition. Upon review of the questionnaire and quadriceps central activation ratio, the study coordinator will determine a subject's eligibility (based on the inclusion and exclusion criteria). We will also collect age, height and weight for all subjects. Participants that qualify will provide written at this time which will be documented by the investigator.

Quadriceps Central Activation Ratio We will use the superimposed burst technique to measure quadriceps muscle strength and to estimate quadriceps activation by calculating the central activation ratio. Subjects will be secured to a chair (Biodex multi-mode dynamometer) with their knees and hips bent to approximately 90 degrees. Subjects will perform a maximal, voluntary isometric knee extension contraction (MVIC) with continuous verbal encouragement from the tester. Once the MVIC reaches a plateau (representing subjects' maximal effort) an electrical stimulus will be manually triggered and delivered directly to the quadriceps through 2 stimulating electrodes which will be secured to the subjects' anterior thigh. The stimulus will cause the quadriceps to twitch resulting in a temporary increase in force production which we will measure. A ratio between the MVIC force and the highest force achieved due to the electrical stimulation will be calculated - this is called the central activation ratio. The electrical stimulus will be delivered manually with a square-wave stimulator in conjunction with a stimulus isolation unit) and will consist of a train of 10 consecutive, square wave pulses of 600 microsecond duration, at an intensity of 125 volts with a carrier frequency of 100 pulses per second. Subjects will have the option of experiencing some "practice" pulses at lower intensity in order to become acclimated to the stimulus and the practice maintaining maximum effort in anticipation of the stimulation.

Randomization Randomization will take place after enrollment and screening take place. The assessor will be blinded in this investigation. Therefore, the clinician responsible for educating patients regarding the exercise protocols will also be responsible for randomization. Randomization will take place on a 1:1 basis. Prior to starting the study, a binary random number generator will be used to generate the randomization scheme. These numbers will then by placed in sealed envelopes and label with individual subject numbers. The randomization envelopes will be stored in a locked drawer and will only be removed by the clinician responsible for randomization. The randomization envelope will then be stored in the participant's research folder.

Quadriceps Hoffmann Reflex We will record muscle reflex activity by delivering a short percutaneous (through the skin) electrical stimulation to femoral nerve located in the inguinal fold. We will measure the reflex response of the quadriceps with surface electromyography. This measure helps to describe the function of a muscle before and after our exercise protocol. Subjects will be positioned comfortably in a lying-down position on a treatment table. Stimuli will be delivered to the femoral nerve by increasing the intensity in small increments with a 10 second rest interval after each stimulus, until the maximum H-reflex amplitude is recorded (Hmax). Then we will increase the stimulus voltage until we obtain a maximum M-wave. The H-reflex represents the proportion of the quadriceps motor neuron pool that is available for voluntary contraction and the M-wave represents the total volume of the quadriceps motor neuron pool and will be used to normalize the H-reflex recordings as H:M ratio. This measurement will be performed bilaterally.

Exercise Intervention Participants in both groups will be instructed on a 14 day exercise (4 supervised session and 10 home sessions) protocol on the day of enrollment. The protocol is comprised of 4 exercises focused on both non-weight bearing and weight bearing quadriceps strengthening. All participants will be asked to complete 3 set of 10 repetitions of isometric quadriceps contractions with a 15 second hold time, supine straight leg raises, body weight squatting, and body weight lunges daily. Participants will be required to complete the single limb exercises on the previously injured limb only. A compliance log will be given to each participant and will be reviewed at each supervised exercise session and at the final study visit. Participants will be instructed to discontinue exercise and contact the principle investigator if they experience knee pain due to the intervention.

Participants in the electromyographic biofeedback supplemented exercise will also be instructed on correct setup and use of the electromyographic biofeedback unit. These instructions will focus on correct placement of the electromyography recording electrodes over quadriceps muscle as well as correct tuning of the feedback threshold for each exercise to maximize the benefit of the intervention. Electromyographic biofeedback will be used during all exercises throughout the course of the study for this group.

Follow-up Testing After 14±1 days of exercise intervention all baseline measures will be re-tested in the same manner as explained above. A supervised exercise session and compliance check will be completed 3±1, 7±1, and 10±1 days following enrollment into the study. No follow-up measurements will be taken at this point, however an exercise compliance log will be collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

* History of primary and uncomplicated knee injury or knee surgery.
* Aged 18-40
* Quadriceps Central Activation Ratio is less than 90%

Exclusion Criteria:

* Currently seeking physical therapy
* Complex knee injury
* Surgical revisions to original procedure
* Pain greater than 4 out of 10 on a visual analog scale at enrollment.
* Active infection
* Current pregnancy
* Cognitive impairment
* Psychiatric disorder requiring daily medication
* Chronic or acute neuropathy
* Known muscular abnormalities
* History of neurological disorders
* History or family history of seizures and/or epilepsy and/or on medications that lower seizure threshold

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kuenze, PhD, Principal Investigator — University of Miami
Locations (1):
- Department of Kinesiology and Sport Sciences, University of Miami, Coral Gables, Florida, United States

REFERENCES:
- [Background] Ng GY, Zhang AQ, Li CK. Biofeedback exercise improved the EMG activity ratio of the medial and lateral vasti muscles in subjects with patellofemoral pain syndrome. J Electromyogr Kinesiol. 2008 Feb;18(1):128-33. doi: 10.1016/j.jelekin.2006.08.010. Epub 2006 Oct 27. PMID 17070701
- [Background] Oravitan M, Avram C. The effectiveness of electromyographic biofeedback as part of a meniscal repair rehabilitation programme. J Sports Sci Med. 2013 Sep 1;12(3):526-32. eCollection 2013. PMID 24149161
- [Background] Christanell F, Hoser C, Huber R, Fink C, Luomajoki H. The influence of electromyographic biofeedback therapy on knee extension following anterior cruciate ligament reconstruction: a randomized controlled trial. Sports Med Arthrosc Rehabil Ther Technol. 2012 Nov 6;4(1):41. doi: 10.1186/1758-2555-4-41. PMID 23126601

RESULTS

PARTICIPANT FLOW:
Groups:
- Electromyographic Biofeedback Group: Participants in the electromyographic biofeedback supplemented exercise will be instructed on correct setup and use of the electromyographic biofeedback unit. Electromyographic biofeedback will be used during all exercises throughout the course of the study for this group. Participants in will be instructed on a 14 day exercise protocol on the day of enrollment. The protocol is comprised of 4 exercises focused on both non-weight bearing and weight bearing quadriceps strengthening. A compliance log will be given to each participant and will be reviewed at each supervised exercise session and at the final study visit. Participants will be instructed to discontinue exercise and contact the principle investigator if they experience knee pain due to the intervention.
  Electromyographic Biofeedback: Electromyographic biofeedback is a device that enables a patient or clinician to measure the intensity of a muscle contraction using electrodes placed on the skin over a muscle of interest.
Period: Overall Study
Arm/Group | Electromyographic Biofeedback Group | Traditional Exercise Group
Started | 2 | 2
Completed | 1 (1 participant dropped out of this study due to the time commitment associated with participation.) | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electromyographic Biofeedback Group | Traditional Exercise Group | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (9.2) | 23.5 (0.7) | 28.5 (7.9)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quadriceps Central Activation Ratio
Description: Subjects will be secured to a chair (Biodex multi-mode dynamometer) with their knees and hips bent to approximately 90-degrees. Subjects will perform a maximal, voluntary isometric knee extension contraction (MVIC) with continuous verbal encouragement from the tester. Once the MVIC reaches a plateau (representing subjects' maximal effort) an electrical stimulus will be manually triggered and delivered directly to the quadriceps through 2 stimulating electrodes which will be secured to the subjects' anterior thigh. The stimulus will cause the quadriceps to twitch resulting in a temporary increase in force production which we will measure. A ratio between the MVIC force and the highest force achieved due to the electrical stimulation will be calculated - this is called the central activation ratio.
Time Frame: Baseline and 14 days
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Electromyographic Biofeedback Group | Traditional Exercise Group
Number analyzed (Participants) | 1 | 2
percentage change from baseline | 15.0 (0) | 20.5 (11.4)

2. Secondary Outcome: Change From Baseline in Quadriceps Hoffmann Reflex
Description: We will record muscle reflex activity by delivering a short percutaneous (through the skin) electrical stimulation to femoral nerve located in the inguinal fold. We will measure the reflex response of the quadriceps with surface electromyography. Subjects will be positioned comfortably in a lying-down position on a treatment table. Stimuli will be delivered to the femoral nerve by increasing the intensity in small increments with a 10-sec rest interval after each stimulus, until the maximum H-reflex amplitude is recorded (Hmax). The H-reflex represents the proportion of the quadriceps motor neuron pool that is available for voluntary contraction and the M-wave represents the total volume of the quadriceps motor neuron pool and will be used to normalize the H-reflex recordings as H:M ratio. This measurement will be performed bilaterally.
Time Frame: Baseline and 14 days
Population: This measure was exclude from the study protocol due to an issue with the equipment utilized to generate the electical pulse. No participants of this study completed the Hoffmann reflex testing protocol at baseline or follow-up visits.
Arm/Group | Electromyographic Biofeedback Group | Traditional Exercise Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data for each individual participant were collected during the time period in which a participant was enrolled in the study (2 weeks). Participants were not subsequently contacted if an adverse event had not been reported during participation.
Arm/Group | Electromyographic Biofeedback Group | Traditional Exercise Group
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No